CLINICAL TRIAL: NCT06417736
Title: Prospective Clinical Study of Fertility-sparing Treatment With a Membrane-inhibiting Formula Combined With Oral Progestins for Endometrial Carcinoma and Hyperplasia in Childbearing-age Women
Brief Title: Prospective Study for Endometrial Carcinoma and Hyperplasia in Childbearing-age Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2023-3614
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Cancer Stage I; Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- membrane-inhibiting formula combined with oral progestins (Experimental): Megestrol acetate(160mg/day) and membrane-inhibiting formula, 24weeks
  Interventions: Drug: Megestrol Acetate 40 MG

INTERVENTIONS:
Drug: Megestrol Acetate 40 MG — 160mg/one time/day
  Other Names: membrane-inhibiting formula

SUMMARY:
The goal of this clinical trial is to evaluate the effect and adverse side effects of membrane-inhibiting formula plus oral progestins as fertility-preserving treatment in patients with early-stage endometrial cancer and endometrial hyperplasia research questions：When taken with oral progestins, does the drug membrane-inhibiting formula shorten the time required for complete endometrial remission? What medical problems do participants have when taking drug membrane-inhibiting formula plus oral progestins? Efficacy, side effects, recurrence, pregnancy, and time to obtain pregnancy in different molecular classifications of POLE-mutated, mismatch repair-deficient(MMRd), p53 wild type(p53wt), and p53-abnormal(p53abn).

Participants will: Take drug membrane-inhibiting formula plus oral progestins every day Visit the clinic once every 3 months for checkups, tests, and hysteroscopy Keep a diary of examination results and pathology

ELIGIBILITY:
Inclusion Criteria:

* 1.18-45 years old with a strong desire to preserve fertility; 2. pathologically diagnosed with primary grade1 or grade2 endometrioid endometrial carcinoma and hyperplasia 3.no signs of suspicious myometrial invasion by enhanced magnetic resonance imaging (MRI) 4. no signs of suspicious extrauterine metastasis by enhanced computed tomography and CT scan of the Lungs

Exclusion Criteria:

* 1.have contraindication for pregnancy. 2.no fertility requiremen 3.have myometrial invasion or extrauterine metastasis 4.pathologically diagnosed with primary grade3 endometrioid endometrial carcinoma or non-endometrioid endometrial carcinoma 5.Any disease or symptom that may affect the implementation of the study or the interpretation of the results

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 75 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
24-week complete response(CR) rate | baseline,12 weeks after treatment,and 24 weeks of treatment
  The treatment response:complete response,no endometrial lesion

SECONDARY OUTCOMES:
36-week CR rate | baseline,12 weeks after treatment,24 weeks of treatment,36 weeks of treatment
  The treatment response:complete response,no endometrial lesion
48-week CR rate | baseline,12 weeks after treatment,24 weeks of treatment,36 weeks of treatment,48 weeks of treatment
  The treatment response:complete response,no endometrial lesion
treatment-related adverse events | baseline,12 weeks after treatment,and 24 weeks of treatment
  analyze the safety of the drug
recurrent rate | baseline,12 weeks after treatment,24 weeks of treatment,36 weeks of treatment,48 weeks of treatment
  cumulative recurrent rate
pregnancy rate | 1-year after CR
  long term fertility results

OTHER OUTCOMES:
CR in different molecular classification | baseline,12 weeks after treatment,24 weeks of treatment,36 weeks of treatment,48 weeks of treatment
  Efficacy in different molecular classification of POLE-mutated, mismatch repair-deficient(MMRd), p53 wild type(p53wt),and p53-abnormal(p53abn)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Doctor, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No